CLINICAL TRIAL: NCT02900547
Title: Blind Assessment of the Concordance Between the Administered Treatment and the Recommendations of a Medical Algorithm Decision Support Software in Systolic Heart Failure
Acronym: PREMEDIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: R2015-15
Record Dates: First submitted 2016-08-12; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-06

CONDITIONS: Hearth Failure, Systolic
Keywords: Systolic Heart Failure; medical algorithm decision support system
MeSH Terms: conditions — Systolic Murmurs; Heart Failure, Systolic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patients with systolic heart failure

SUMMARY:
The PREMEDIC is a prospective, observational study. Patients hospitalized for Systolic Heart Failure will be enrolled and health data will be collected at hospital admission and during hospital stay. No data will be collected before detailed information is given to the patient and a non-opposition is obtained.

The aim of this observational and prospective study is to evaluate the concordance actual patient management during the in hospital treatment of heart failure and the therapeutic proposals from a medical algorithmic decision support software.

DETAILED DESCRIPTION:
Main Objective:

The aim of this observational and prospective study is to evaluate retrospectively the concordance between the actual systolic heart failure patient management during the inhospital treatment of heart failure (as recorded from the usual healthcare data collected) and the therapeutic proposals from a medical algorithmic decision support software.

Secondary Objectives:

To study the evolution of biological, hepatic and cardiopulmonary ultrasound usual markers in hospitalization, in connection with the duration of hospitalization and drug administered.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or over
* Patients hospitalized for decompensated systolic heart failure
* Patients informed

Exclusion Criteria:

* Patients unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for acutely decompensated systolic heart failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Retrospective evaluation of the concordance between the drug therapy actually used and the therapeutic algorithm's proposals | an average of 7 days

SECONDARY OUTCOMES:
Duration of hospitalization (number of days) | an average of 7 days
Weight evolution (Kilograms) | an average of 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France